CLINICAL TRIAL: NCT01257568
Title: A Prospective, Post-market, Multi-center Study of the Outcomes of the Rejuvenate® Modular Hip System
Brief Title: Rejuvenate Modular Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rejuvenate Modular Hip System (Other): Rejuvenate Modular Hip
  Interventions: Device: Rejuvenate Modular Hip

INTERVENTIONS:
Device: Rejuvenate Modular Hip — Rejuvenate Modular Hip

SUMMARY:
This study will be an evaluation of the Rejuvenate® Modular Hip System for primary total hip replacement (THR) with a cementless application in a consecutive series of patients who meet the eligibility criteria. Subjects will be evaluated for freedom of hip revision at 5 years and clinical outcomes for up to 10 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed an IRB approved, study specific Informed Patient Consent Form.
* Patient is a male or non-pregnant female age 18 years or older at time of study device implantation.
* Patient has primary diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD).
* Patient is a candidate for a primary cementless total hip replacement.
* Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.
* Patient's operative femur templates to Rejuvenate® Modular Stem size 7-12.

Exclusion Criteria:

* Patient has a Body Mass Index (BMI) ≥ 40.
* Patient has an active or suspected latent infection in or about the affected hip joint at time of study device implantation.
* Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.
* Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's Disease) leading to progressive bone deterioration.
* Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
* Patient requires revision surgery of a previously implanted total hip replacement or hip fusion to the affected joint.
* Patient has a known sensitivity to device materials.
* Patient is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-11; Primary Completion 2017-06-06 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh Mittal, M.D., Principal Investigator — The Orthopedic Center; Joseph Nessler, M.D., Principal Investigator — St. Cloud Orthopaedic Associates; Lawrence Morawa, M.D., Principal Investigator — Oakwood Healthcare System
Locations (3):
- United States (3):
  - Oakwood Healthcare, Dearborn, Michigan
  - St. Cloud Orthopaedics Associates, Sartell, Minnesota
  - The Orthopedic Center, Tulsa, Oklahoma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in the Rejuvenate Modular Hip Stem study was terminated early. Participants can have one or both hips replaced. If both hips were enrolled in the study and only one hip completed the primary endpoint the participant is counted as completed.
Pre-assignment Details: 42 participants/44 hips - 2 participants/2 hips censored = 40 participants/42 hips followed. There were 25 revisions, but one bilateral participant had one hip revised and the other hip completed the primary endpoint, this participant is counted as completed and not in the revision category.
Units Other Than Participants: Hips
Groups:
- Rejuvenate Modular Hip System: Participants who received the Rejuvenate Modular stem/neck can have one or both hips replaced. If both hips were replaced, but one hip completed the primary endpoint, the participant is counted as completed.
Period: Overall Study
Arm/Group | Rejuvenate Modular Hip System
Started | 40; 42 Hips
Completed | 7; 9 Hips
Not Completed | 33; 33 Hips
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 6
Not completed — Terminated | 1
Not completed — Component Revision | 24

BASELINE CHARACTERISTICS:
Population: Includes all participants who received the Rejuvenate Modular neck/stem and were not censored from analysis.
Units Other Than Participants: Hips
Groups:
- Rejuvenate Modular Hip System: All subjects who received the Rejuvenate Modular stem/neck.
Arm/Group | Rejuvenate Modular Hip System
Number analyzed (Participants) | 40
Number analyzed (Hips) | 42
Age, Continuous [Mean (Full Range); unit: years] — For bilateral participants, age at the time of surgery for the first hip enrolled is used for the baseline measurement
  years
    Age | 62.50 [46 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate of the Rejuvenate Modular Stem/Neck
Description: The success rate is defined as freedom from Rejuvenate Modular femoral stem/neck construct revision/removal for any reason.
Time Frame: 5 years postoperative
Measure: Number; unit: Surviving Hips
Units Other Than Participants: Hips
Arm/Group | Rejuvenate Modular Hip System
Number analyzed (Participants) | 40
Number analyzed (Hips) | 42
Surviving Hips | 8

2. Secondary Outcome: Biomechanical Measurement of Femoral Offset
Description: Change from Preoperative Natural Femoral Offset to Postoperative Femoral Offset at 6-weeks postoperative measured in millimeters.
Time Frame: 6 weeks
Population: The data presented on these 41 hips is likely inaccurate due to issues and variations in data collection.
Measure: Median (Inter-Quartile Range); unit: mm
Units Other Than Participants: Hips
Arm/Group | Rejuvenate Modular Hip System
Number analyzed (Participants) | 39
Number analyzed (Hips) | 41
mm | -2 [-41 to 4]

3. Secondary Outcome: Biomechanical Measurement of the Vertical Distance of the Planned Hip Center of Rotation
Description: Change from preoperative vertical distance of the anatomic hip center to the planned center of rotation of the hip to the postoperative distance from the planned center of rotation at 6 weeks measured in millimeters.
Time Frame: 6 weeks
Population: The data presented on these 5 hips is likely inaccurate due to issues and variations in data collection.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Rejuvenate Modular Hip System
Number analyzed (Participants) | 5
mm | -4 [-38 to 1]

4. Secondary Outcome: Biomechanical Measurement of the Horizontal Distance of the Planned Hip Center of Rotation
Description: Change from preoperative horizontal distance of the anatomic hip center to the planned center of rotation of the hip to the postoperative distance from the planned center of rotation at 6 weeks measured in millimeters.
Time Frame: 6 weeks
Population: The data presented on these 5 hips is likely inaccurate due to issues and variations in data collection.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Rejuvenate Modular Hip System
Number analyzed (Participants) | 5
mm | 0 [-2 to 2]

5. Secondary Outcome: Mean Harris Hip Score at Each Visit
Description: The Harris Hip Score (HHS) assesses pain, function, joint deformity and range of motion. Scores can range from 0 to 100 with 0 being the worst and 100 being the best score. A score of 80-100 is considered good-excellent and a score of less than or equal to 79 is considered fair-poor.
  90-100 = excellent 80-89 = good 70-79 = fair 0-69 = poor
Time Frame: pre-op, 6 wk, 1, 2, 3, 4, 5, 7 year
Population: Participants/hips with available data. Overall number of participants and units analyzed is based upon the preoperative population.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Groups:
- Rejuvenate Modular Hip System: Participants who received the Rejuvenate Modular stem/neck.
Arm/Group | Rejuvenate Modular Hip System
Number analyzed (Participants) | 40
Number analyzed (Hips) | 42
units on a scale
  HHS Mean Preoperative Score | 55.48 (9.88)
  HHS Mean 6 Week Score: number analyzed (Participants) | 39
  HHS Mean 6 Week Score: number analyzed (Hips) | 41
  HHS Mean 6 Week Score | 69.88 (12.97)
  HHS Mean 1 Year Score: number analyzed (Participants) | 34
  HHS Mean 1 Year Score: number analyzed (Hips) | 36
  HHS Mean 1 Year Score | 94.25 (7.65)
  HHS Mean 2 Year Score: number analyzed (Participants) | 22
  HHS Mean 2 Year Score: number analyzed (Hips) | 24
  HHS Mean 2 Year Score | 89.92 (11.49)
  HHS Mean 3 Year Score: number analyzed (Participants) | 16
  HHS Mean 3 Year Score: number analyzed (Hips) | 18
  HHS Mean 3 Year Score | 90.83 (11.71)
  HHS Mean 4 Year Score: number analyzed (Participants) | 10
  HHS Mean 4 Year Score: number analyzed (Hips) | 11
  HHS Mean 4 Year Score | 90.82 (15.65)
  HHS Mean 5 Year Score: number analyzed (Participants) | 7
  HHS Mean 5 Year Score: number analyzed (Hips) | 8
  HHS Mean 5 Year Score | 97.88 (2.1)
  HHS Mean 7 Year Score: number analyzed (Participants) | 4
  HHS Mean 7 Year Score: number analyzed (Hips) | 5
  HHS Mean 7 Year Score | 96.00 (7.38)

6. Secondary Outcome: Mean SF-12 Scores at Each Visit
Description: The SF-12 Health Survey is a 12-item patient completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: pre-op, 6 wk, 1, 2, 3, 4, 5, 7 year
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | Rejuvenate Modular Hip System
Number analyzed (Participants) | 40
Number analyzed (Hips) | 42
units on a scale
  Mean SF-12 Physical Score Preoperative | 33.26 (8.33)
  Mean SF-12 Physical Score 6 weeks | 37.07 (7.72)
  Mean SF-12 Physical Score 1 year: number analyzed (Participants) | 31
  Mean SF-12 Physical Score 1 year: number analyzed (Hips) | 33
  Mean SF-12 Physical Score 1 year | 51.98 (7.34)
  Mean SF-12 Physical Score 2 years: number analyzed (Participants) | 11
  Mean SF-12 Physical Score 2 years: number analyzed (Hips) | 11
  Mean SF-12 Physical Score 2 years | 46.83 (12.06)
  Mean SF-12 Physical Score 3 years: number analyzed (Participants) | 10
  Mean SF-12 Physical Score 3 years: number analyzed (Hips) | 11
  Mean SF-12 Physical Score 3 years | 50.15 (9.3)
  Mean SF-12 Physical Score 4 years: number analyzed (Participants) | 6
  Mean SF-12 Physical Score 4 years: number analyzed (Hips) | 7
  Mean SF-12 Physical Score 4 years | 49.04 (10.55)
  Mean SF-12 Physical Score 5 years: number analyzed (Participants) | 5
  Mean SF-12 Physical Score 5 years: number analyzed (Hips) | 6
  Mean SF-12 Physical Score 5 years | 53.61 (5.4)
  Mean SF-12 Physical Score 7 years: number analyzed (Participants) | 4
  Mean SF-12 Physical Score 7 years: number analyzed (Hips) | 4
  Mean SF-12 Physical Score 7 years | 48.86 (5.62)
  Mean SF-12 Mental Score Preoperative | 51.6 (13.48)
  Mean SF-12 Mental Score 6 weeks | 54.35 (9.37)
  Mean SF-12 Mental Score 1 year: number analyzed (Participants) | 31
  Mean SF-12 Mental Score 1 year: number analyzed (Hips) | 33
  Mean SF-12 Mental Score 1 year | 55.01 (9.26)
  Mean SF-12 Mental Score 2 years: number analyzed (Participants) | 11
  Mean SF-12 Mental Score 2 years: number analyzed (Hips) | 11
  Mean SF-12 Mental Score 2 years | 53.99 (10.13)
  Mean SF-12 Mental Score 3 years: number analyzed (Participants) | 10
  Mean SF-12 Mental Score 3 years: number analyzed (Hips) | 11
  Mean SF-12 Mental Score 3 years | 54.47 (10.03)
  Mean SF-12 Mental Score 4 years: number analyzed (Participants) | 6
  Mean SF-12 Mental Score 4 years: number analyzed (Hips) | 7
  Mean SF-12 Mental Score 4 years | 48.77 (10.99)
  Mean SF-12 Mental Score 5 years: number analyzed (Participants) | 5
  Mean SF-12 Mental Score 5 years: number analyzed (Hips) | 6
  Mean SF-12 Mental Score 5 years | 55.62 (6.88)
  Mean SF-12 Mental Score 7 years: number analyzed (Participants) | 4
  Mean SF-12 Mental Score 7 years: number analyzed (Hips) | 4
  Mean SF-12 Mental Score 7 years | 58.84 (2.68)

7. Secondary Outcome: Mean Lower Extremity Activity Scale (LEAS) Scores at Each Visit
Description: The LEAS is completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level.
Time Frame: pre-op, 6 wk, 1, 2, 3, 4, 5, 7 year
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Arm/Group | Rejuvenate Modular Hip System
Number analyzed (Participants) | 40
Number analyzed (Hips) | 42
units on a scale
  Mean LEAS Score Preoperative | 8.88 (2.58)
  Mean LEAS Score 6 weeks | 7.45 (1.53)
  Mean LEAS Score 1 year: number analyzed (Participants) | 32
  Mean LEAS Score 1 year: number analyzed (Hips) | 34
  Mean LEAS Score 1 year | 11.32 (3.05)
  Mean LEAS Score 2 years: number analyzed (Participants) | 11
  Mean LEAS Score 2 years: number analyzed (Hips) | 11
  Mean LEAS Score 2 years | 11.18 (3.06)
  Mean LEAS Score 3 years: number analyzed (Participants) | 11
  Mean LEAS Score 3 years: number analyzed (Hips) | 13
  Mean LEAS Score 3 years | 11.85 (2.76)
  Mean LEAS Score 4 years: number analyzed (Participants) | 6
  Mean LEAS Score 4 years: number analyzed (Hips) | 7
  Mean LEAS Score 4 years | 11.29 (2.93)
  Mean LEAS Score 5 years: number analyzed (Participants) | 5
  Mean LEAS Score 5 years: number analyzed (Hips) | 6
  Mean LEAS Score 5 years | 13.33 (3.14)
  Mean LEAS Score 7 years: number analyzed (Participants) | 4
  Mean LEAS Score 7 years: number analyzed (Hips) | 5
  Mean LEAS Score 7 years | 11.60 (1.14)

8. Secondary Outcome: Occurrence of Subsidence at Six Weeks, Stem Migration, Unstable Fixation and Radiographic Instability (Radiolucency)
Description: Radiographic stability of the stem is defined as having the following: no radiographic indication of progressive radiolucent lines greater than or equal to 2 mm around the entire femoral component, and no radiographic indication of progressive subsidence of the femoral component of great than or equal to 5 mm. Only subsidence was measured at 6 weeks, migration and fixation are analyzed beginning at 1 year postoperative.
Time Frame: 6 wks,1,2,3,4,5 yrs
Population: Participants/hips with available data. Overall number of participants and units analyzed is based upon the preoperative population. The number of hips analyzed for stem subsidence equals the number of cases with a readable AP Femur or Pelvis x-ray.
Measure: Number; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Rejuvenate Modular Hip System
Number analyzed (Participants) | 40
Number analyzed (Hips) | 42
Hips
  Stem Subsidence-6 weeks | 5
  Stem Migration-1 year: number analyzed (Participants) | 33
  Stem Migration-1 year: number analyzed (Hips) | 35
  Stem Migration-1 year | 4
  Stem Migration-2 years: number analyzed (Participants) | 20
  Stem Migration-2 years: number analyzed (Hips) | 20
  Stem Migration-2 years | 4
  Stem Migration-3 years: number analyzed (Participants) | 14
  Stem Migration-3 years: number analyzed (Hips) | 15
  Stem Migration-3 years | 6
  Stem Migration-4 years: number analyzed (Participants) | 9
  Stem Migration-4 years: number analyzed (Hips) | 9
  Stem Migration-4 years | 4
  Stem Migration-5 years: number analyzed (Participants) | 3
  Stem Migration-5 years: number analyzed (Hips) | 3
  Stem Migration-5 years | 0
  Stem Fixation Unstable-1 year: number analyzed (Participants) | 33
  Stem Fixation Unstable-1 year: number analyzed (Hips) | 35
  Stem Fixation Unstable-1 year | 1
  Stem Fixation Unstable-2 years: number analyzed (Participants) | 21
  Stem Fixation Unstable-2 years: number analyzed (Hips) | 23
  Stem Fixation Unstable-2 years | 1
  Stem Fixation Unstable-3 years: number analyzed (Participants) | 15
  Stem Fixation Unstable-3 years: number analyzed (Hips) | 17
  Stem Fixation Unstable-3 years | 0
  Stem Fixation Unstable-4 years: number analyzed (Participants) | 9
  Stem Fixation Unstable-4 years: number analyzed (Hips) | 10
  Stem Fixation Unstable-4 years | 0
  Stem Fixation Unstable-5 years: number analyzed (Participants) | 4
  Stem Fixation Unstable-5 years: number analyzed (Hips) | 4
  Stem Fixation Unstable-5 years | 0
  Radiographic stability-6 weeks | 42
  Radiographic stability-1 year: number analyzed (Participants) | 33
  Radiographic stability-1 year: number analyzed (Hips) | 35
  Radiographic stability-1 year | 35
  Radiographic stability-2 years: number analyzed (Participants) | 19
  Radiographic stability-2 years: number analyzed (Hips) | 20
  Radiographic stability-2 years | 20
  Radiographic stability-3 years: number analyzed (Participants) | 15
  Radiographic stability-3 years: number analyzed (Hips) | 17
  Radiographic stability-3 years | 17
  Radiographic stability-4 years: number analyzed (Participants) | 8
  Radiographic stability-4 years: number analyzed (Hips) | 9
  Radiographic stability-4 years | 9
  Radiographic stability-5 years: number analyzed (Participants) | 4
  Radiographic stability-5 years: number analyzed (Hips) | 4
  Radiographic stability-5 years | 4

ADVERSE EVENTS:
Time Frame: To 10 years postoperative. All AEs that meet the definition of serious, excluding elective procedures, and all AEs related to the operative site, regardless of seriousness.
Description: Censored were not included as at risk.
Groups:
- Operative Adverse Events: Rejuvenate Modular Stem/Neck. Operative site events are reported by hip because in the case of bilateral participants (this is when one participant has both hips enrolled in the study), an event can occur in one hip, both hips or the same hip at different times and are counted separately for this reason.
- Non-Operative Adverse Events: Rejuvenate Modular Stem/Neck. Non-operative site events are reported by participant.
Arm/Group | Operative Adverse Events | Non-Operative Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 25/42 | 4/40
Other Adverse Events (participants affected / at risk) | 9/42 | 7/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Adverse Events (N=42) | Non-Operative Adverse Events (N=40)
Operative Site (Infections and infestations) | 1 (1) | 0/0 (0)
Operative Site (Injury, poisoning and procedural complications) | 1 (1) | 0/0 (0)
Operative Site (Musculoskeletal and connective tissue disorders) | 3 (3) | 0/0 (0)
Operative Site (Product Issues) | 22 (22) | 0/0 (0)
Systemic Event (Cardiac disorders) | 0/0 (0) | 1 (1)
Systemic Event (Gastrointestinal disorders) | 0/0 (0) | 1 (1)
Systemic Event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 1 (1)
Systemic Event (Nervous system disorders) | 0/0 (0) | 1 (1)
Systemic Event (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Adverse Events (N=42) | Non-Operative Adverse Events (N=40)
Operative Site (Musculoskeletal and connective tissue disorders) | 6 (6) | 0/0 (0)
Operative Event (Product Issues) | 4 (5) | 0/0 (0)
Systemic Events (Product Issues) | 0/0 (0) | 7 (7)

LIMITATIONS AND CAVEATS:
Primary Outcome Note: Due to the large number of terminations and halting enrollment early in the study, the primary endpoint analysis will not be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator shall have privileges for their own center's results. These manuscripts and abstracts will be delayed until after the 5-year multi-center publication is submitted. All publications shall be submitted to the sponsor for review at least 60 days prior to submission for publication. The sponsor shall not edit or otherwise influence the publications other than to ensure that confidential information is not disclosed and that the data is accurately represented.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2009-10-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT01257568/Prot_SAP_ICF_000.pdf